CLINICAL TRIAL: NCT04584398
Title: Effect of Respiratory Training and Steam Inhalation With WellO2 Device on Lung Function and Respiratory Symptoms in Patients With Chronic Obstructive Lung Diseases - a Pilot Study
Brief Title: Effects of Combined Respiratory Muscle Training and Steam Inhalation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: WellO2 Oy (Industry)
Collaborators: Oy Medfiles (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HA010
Record Dates: First submitted 2020-09-21; First posted 2020-10-14 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-09

CONDITIONS: Airway Obstruction; Asthma; COPD
Keywords: Respiration; Respiratory muscle training; Steam inhalation
MeSH Terms: conditions — Airway Obstruction; Asthma; Pulmonary Disease, Chronic Obstructive; Respiratory Aspiration | interventions — Breathing Exercises

STUDY DESIGN:
Intervention Model Description: Randomized, controlled, single-blind parallel design with 50-60 subjects suffering from obstructive diseases such as asthma or COPD or both.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The study is conducted as a randomized, single-blind (for evaluators), controlled, 30 days intervention trial with two parallel groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The intervention group (A) will perform respiratory muscle training and steam inhalation with WellO2 device for 30 days.
  Interventions: Device: Respiratory muscle training with steam inhalation
- Control (No Intervention): The control group (B) will continue on their conventional treatment without respiratory muscle training or steam inhalation with WellO2. After 30 days, the group B performs the same 30-day intervention with the WellO2 device (test) as the group A.

INTERVENTIONS:
Device: Respiratory muscle training with steam inhalation
  Arms: Intervention

SUMMARY:
The purpose of this investigation is to obtain more information on the efficacy and safety of respiratory training methods with WellO2 in patients with asthma and COPD. Such a training may offer an additional, non-pharmacological way for treatment and therapy of asthma and COPD.

DETAILED DESCRIPTION:
Numerous respiratory muscle training (RMT) experiments with healthy subjects, as well as with patients of chronic obstructive pulmonary disease (COPD), bronchiectasis and asthma, have been reported since 80's. Respiratory training with WellO2 device was used in a clinical pilot study by Huttunen and Rantala to investigate effects of steam inhalation and RMT on voice quality in patients with voice symptoms. No adverse effects were found in that study.

The present study is designed to investigate further the RMT and steam inhalation on lung function and respiratory symptoms with subjects suffering from obstructive diseases such as asthma and COPD. The results may be used later in statistical power calculations and to determine the endpoints of larger clinical trial with the investigational device.

Asthma is still an increasing problem in many countries, even though, incidence of the most severe asthma cases is in decline due to earlier diagnosis, better control and earlier intervention practices. The prevalence of asthma and COPD in western countries is around 10 % and 5 %, respectively. The prevalence of COPD is higher in the countries where smoking and poor quality of inhaled air are common.

The treatment of asthma is based on treatment of eosinophilic inflammation of the airways by inhaled corticosteroids and on treatment of bronchoconstriction by sympathomimetic bronchodilators, short-acting and long-acting. The drugs may, however, induce side effects like voice disorders and cardiac symptoms (palpitation, tachycardia and extrasystoles).

Therefore, in many cases the doses of the drugs cannot continuously be kept at the highest effective level. Therefore, non-pharmacological methods can complement the treatment portfolio. The breathing physiotherapy by respiratory muscle training and warm steam inhalation can offer an additive treatment method for patients with airway obstruction.

It is possible that training with the combination of positive counter pressure and steam inhalation methods can induce significant improvement in ventilatory function variables and respiratory symptoms in asthmatics who have kept their ordinary pharmacological therapy at a constant level. Based on the previous scientific evidence found on the public domains, it can be expected that the respiratory muscle strength will be increased offering a possibility for more effective pulmonary mechanics, ventilation and lung volumes. In addition, exhaling against resistance will induce a positive end expiratory pressure (PEEP) effect which can open narrowed airways and make the distribution of alveolar ventilation less heterogeneous. This can improve gas exchange in the lungs and increase the level of low oxygen saturation in arterial blood.

In COPD, drugs can improve the airway changes, irreversible thickening of the airway walls, and chronic inflammation only partially. Therefore, breathing physiotherapy may offer an additive method to improve lung function and gas exchange, and to diminish dyspnoea and other symptoms like cough. The mechanisms of RMT are principally the same in asthma and COPD. Patients with obstructive airway disease frequently have both COPD and asthma, partly reversible or irreversible.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent
2. Age 18-65 years
3. Ethnic origin: Finnish
4. Both men and women are included
5. Diagnosed COPD or asthma or both
6. The duration of the illness at least 1 year, and the disease is at a stable stage
7. Pulmonary medication: unchanged for 4 weeks before the start of the study and throughout the study
8. Severity of the disease: mild, moderate or severe
9. The baseline FEV1 45-90 % of predicted normal value (Kainu et al 2016)
10. Eventual previous smoking has been ceased at least four weeks before the study
11. Compliance and commitment to the study (volunteered study subjects)

Exclusion Criteria:

1. Previous history of pneumothorax
2. Unstable emphysema
3. Chest, abdominal, or cerebral aneurysms
4. Epilepsy
5. Chronic nose bleeding
6. Recent (< 3 months) surgical operations
7. Pregnancy
8. Unstable mental health issues
9. Alcohol consumption more than 10 portions/week (one portion is e.g. 4 cl of strong drinks including 40 % alcohol by volume)
10. Drug addiction
11. Non-compliance to the study protocol
12. History of worsening asthma symptoms at sauna
13. Any other pulmonary disease than asthma or COPD
14. Any other major illnesses such as heart failure, coronary artery disease, neurological diseases or type 1 diabetes
15. Smoking during the study period of 16 weeks

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2021-03-02 (Estimated); Study Completion 2021-03-30 (Estimated)

PRIMARY OUTCOMES:
Change in forced expiratory volume in one second (FEV1) measured with spirometry | 30 days intervention plus 190 days washout period
  Statistical difference of FEV1 between and within the arms compared to the baseline

SECONDARY OUTCOMES:
Change in vital capacity (VC) measured with spirometry | 30 days intervention plus 190 days washout period
  Statistical difference between and within the arms compared to the baseline
Change in forced vital capacity (FVC) measured with spirometry | 30 days intervention plus 190 days washout period
  Statistical difference between and within the arms compared to the baseline
Change in peak expiratory flow (PEF) measured with spirometry | 30 days intervention plus 190 days washout period
  Statistical difference between and within the arms compared to the baseline
Change in forced expiratory volume in one second / vital capacity (FEV1/VC) measured with spirometry | 30 days intervention plus 190 days washout period
  Statistical difference between and within the arms compared to the baseline
Change in forced expiratory volume in one second / forced vital capacity (FEV1/FVC) measured with spirometry | 30 days intervention plus 190 days washout period
  Statistical difference between and within the arms compared to the baseline
Change in maximum expiratory flow at 50% of FVC (MEF50) measured with spirometry | 30 days intervention plus 190 days washout period
  Statistical difference between and within the arms compared to the baseline
Change in maximal mid-expiratory flow (MMEF) measured with spirometry | 30 days intervention plus 190 days washout period
  Statistical difference between and within the arms compared to the baseline
Bronchodilatation test with inhaled salbutamol (0,4 mg) | 30 days intervention plus 190 days washout period
  Statistical difference between and within the arms compared to the baseline
Change in arterial oxygen saturation SpO2 (%) | 30 days intervention plus 190 days washout period
  Statistical difference between and within the arms compared to the baseline
Change in maximal expiratory and inspiratory airway pressures (MEP and MIP) | 30 days intervention plus 190 days washout period
  Statistical difference between and within the arms compared to the baseline
Change in systolic and diastolic blood pressure at rest | 30 days intervention plus 190 days washout period
  Statistical difference between and within the arms compared to the baseline
Change in heart rate at rest | 30 days intervention plus 190 days washout period
  Statistical difference between and within the arms compared to the baseline

OTHER OUTCOMES:
Adverse events | 120 days
  Total number and severity of adverse events between the test and control group during the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Jukka Heinijoki, MD, Principal Investigator — Medical center Johanneksen Klinikka
Locations (1):
- Medical Center Johanneksen Klinikka, Tampere, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Manufacturer's web address — http://www.wello2.com